CLINICAL TRIAL: NCT05778760
Title: Prospective, Double-Blinded, Randomized Head-to-Head Study of Topical Adapinoid Versus Topical Retinol
Brief Title: Prospective Study of Topical Adapinoid Versus Topical Retinol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Actera (Sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADAP_RET
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Wrinkle
Keywords: anti-aging; skin care
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinol (Active Comparator): Product will be used once daily in the evening for 12 weeks. 1-2 pumps (size of quarter) of product will be applied on the face.
  Interventions: Other: Retinol
- Adapinoid (Experimental): Product will be used once daily in the evening for 12 weeks. 1-2 pumps (size of quarter) of product will be applied on the face.
  Interventions: Other: Adapinoid

INTERVENTIONS:
Other: Retinol — Topical retinol (0.5%) applied to the face
  Arms: Retinol
Other: Adapinoid — Topical Adapinoid (0.5%) applied to the face
  Arms: Adapinoid

SUMMARY:
This study is to analyze and compare the effects of applying two topical vitamin-A derived ingredients on facial skin health, appearance and tolerability. One of these ingredients is retinol, and the other is Adapinoid, also known as Oleyl Adapalenate, a novel anti-aging ingredient.

DETAILED DESCRIPTION:
We want to assess the effect of applying vitamin A-derived ingredients on facial skin health, appearance, and tolerability. One of these ingredients is retinol, and the other is Adapinoid, also known as Oleyl Adapalenate.

In this study, participants will be randomized to either receiving a retinol product, or an Adapinoid product and they will be assessed at three follow up visits at week 4, week 8, and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 35 years old and 65 years old

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Subjects using any topical retinoid, acetyl zingerone, vitamin C, bakuchiol, hyaluronic acid or benzoyl peroxide containing topical product within 2 weeks of starting study or any subject unwilling to refrain from washout prior to enrollment.
* Subjects with any of the following facial cosmetic treatments in the past 3 months or those who are unwilling to withhold the following facial cosmetic treatments during study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Facial fine lines and wrinkles | 12 weeks
  Change in severity of fine lines and wrinkles measured by photographic analysis (BTBP 3D Camera System)

SECONDARY OUTCOMES:
Facial fine lines and wrinkles | 4 weeks
  Change in severity of fine lines and wrinkles measured by photographic analysis (BTBP 3D Camera System)
Facial fine lines and wrinkles | 8 weeks
  Change in severity of fine lines and wrinkles measured by photographic analysis (BTBP 3D Camera System)
Skin redness | 4 weeks
  Change in the appearance of skin redness measured by photographic analysis (BTBP 3D Camera System)
Skin redness | 8 weeks
  Change in the appearance of skin redness measured by photographic analysis (BTBP 3D Camera System)
Skin redness | 12 weeks
  Change in the appearance of skin redness measured by photographic analysis (BTBP 3D Camera System)
Facial skin pigment evenness | 4 weeks
  Change in the appearance of facial skin pigment intensity measured by photographic analysis (BTBP 3D Camera System)
Facial skin pigment evenness | 8 weeks
  Change in the appearance of facial skin pigment intensity measured by photographic analysis (BTBP 3D Camera System)
Facial skin pigment evenness | 12 weeks
  Change in the appearance of facial skin pigment intensity measured by photographic analysis (BTBP 3D Camera System)
Self-perception of skin health and appearance | 4 weeks
  Survey-based self-assessment of aspects of skin health and appearance
Self-perception of skin health and appearance | 8 weeks
  Survey-based self-assessment of aspects of skin health and appearance
Self-perception of skin health and appearance | 12 weeks
  Survey-based self-assessment of aspects of skin health and appearance
Tolerability of product | 4 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin product
Tolerability of product | 8 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin product
Tolerability of product | 12 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin product

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen N, Afzal N, Min M, Ahmad N, Afzal L, Burney W, Chambers CJ, Sivamani RK. A prospective, double-blinded, randomized head-to-head clinical trial of topical adapinoid (oleyl adapalenate) versus retinol. Skin Health Dis. 2024 Nov 4;4(6):e469. doi: 10.1002/ski2.469. eCollection 2024 Dec. PMID 39624736